CLINICAL TRIAL: NCT04472468
Title: Primary Percutaneous Pericardiotomy for Malignant Pericardial Effusion (PMAP) - a Randomized Study
Brief Title: Primary Percutaneous Pericardiotomy for Malignant Pericardial Effusion (PMAP)
Acronym: PMAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slower than target enrollment.
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, GuangMing Tan, Honorary Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C18-004
Record Dates: First submitted 2020-07-13; First posted 2020-07-15 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Pericardial Effusion Malignant
Keywords: pericardial effusion, malignancy, pericardiotomy.
MeSH Terms: conditions — Pericardial Effusion; Neoplasms

STUDY DESIGN:
Intervention Model Description: multi-center, randomized, prospective, open label controlled pragmatic trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (pericardiotomy) (Experimental): * Patient in this arm will receive balloon pericardiotomy before insertion of pericardiocentesis.
  * An 20mm over-the-wire ultra-non-compliant Percutaneous Transluminal Angioplasty Balloon is used to dilate the pericardium.
  * Success of balloon pericardiotomy is confirmed by full inflation of the balloon which is confirmed on two orthogonal projections.
  * Standard pericardiocentesis with prolonged drainage is performed afterwards.
  * Pericardial drain is removed when output is less than 100cc/day
  Interventions: Device: Percutaneous Balloon Pericardiotomy
- Control (standard pericardiocentesis) (No Intervention): * Standard pericardiocentesis procedure is performed using standard pigtail pericardial drain. - Pericardial fluid is then tapped until dry on table.
  * Pericardial drain is removed when output is less than 100cc/day

INTERVENTIONS:
Device: Percutaneous Balloon Pericardiotomy — * Subxiphoid approach under fluoroscopic guidance is used.
  * An 20mm over-the-wire ultra-non-compliant Percutaneous Transluminal Angioplasty Balloon is advanced into the pericardial space.
  * Success of balloon pericardiotomy is confirmed by full inflation of the balloon which is confirmed on two orthogonal projections.
  Other Names: balloon pericardiotomy
  Arms: Treatment (pericardiotomy)

SUMMARY:
Pericardial effusion is a common complication in patients with metastatic malignancy. While pericardiocentesis provide effective relieve from life-threatening situation such as cardiac tamponade, recurrence of pericardial effusion after pericardiocentesis is common. We hypothesize that percutaneous balloon pericardiotomy in addition to standard pericardiocentesis with prolonged drainage can prevent pericardial effusion recurrence in patients with malignant pericardial effusion.

DETAILED DESCRIPTION:
Pericardial effusion is a common complication in patients with metastatic malignancy with an incidence as high as 21%. The occurrence of malignant pericardial effusion significantly impacts on patient's survival and quality of life. While pericardiocentesis provide effective relieve from life-threatening situation such as cardiac tamponade, recurrence of pericardial effusion after pericardiocentesis is common and occurs in as high as 31% of patients. Retrospective data has shown that prolonged pericardial drainage might reduce the recurrence rate but at the cost of increased risk of infection and prolonged hospital stay. Surgical pericardiotomy was used in the past but was not shown to reduce recurrence over prolonged pericardial drainage and is associated with a higher rate of complications. Surgical pericardial window creation via a mini-thoracotomy might be an effective treatment and can be considered in patient with pericardial tamponade. The safety and feasibility of Percutaneous Balloon pericardiotomy (PBP) has been first described 1993 and has been shown to be an alternative treatment for patient with malignant pericardial effusion. However, no data is available on the efficacy of PBP in reducing the recurrence of pericardial effusion, in comparison with standard pericardiocentesis with prolonged drainage. We aim to perform a single centre, randomized, prospective, open label controlled pragmatic trial to compare percutaneous balloon pericardiotomy (treatment) to standard pericardiocentesis with prolonged drainage (control) in preventing pericardial effusion recurrence in patients with malignant pericardial effusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed active malignancy AND,
* Presence of at least moderate (>10cm) pericardial effusion on CT or Echocardiography

Exclusion Criteria:

* Patients unable to give an informed consent,
* Previous history of open-heart surgery
* Previous history of pericardial window or pericardial instillation of sclerosing therapy.
* Scheduled thoracic or cardiac surgery within the next 3 months
* Patients with contraindications for endovascular procedure such as disseminated intravascular coagulopathy or significant ongoing bleeding tendency, and systemic septicaemia.
* Patient with small or loculated pericardial effusion that is not accessible by subxiphoid approach.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Pericardial effusion recurrence | 3 months
  Recurrence of pericardial effusion after index procedure, defined as development of moderate or more pericardial effusion (>10mm) on follow-up imaging.
Procedural related complications | Immediate after intervention
  Procedural related complications including procedural related death, need for urgent surgical intervention, pleural effusion and pneumothorax

SECONDARY OUTCOMES:
Survival | 3 months
  overall survival
Pericardial effusion free survival | 3 months
  survival without recurrence of pericardial effusion
cardiac tamponade | 3 months
  Occurrence of cardiac tamponade as defined by echocardiographic finding of any of the following: 1. diastolic collapse of the right atrium, 2. Diastolic collapse of the right ventricle, 3. respiratory variation of the mitral E' velocity > 25% or tricuspid E' velocity >40%, 4. dilated IVC >20mm and <50% respiratory reduction.
Quality of life measure (using Functional Assessment of Cancer Therapy - General version (Chinese version)). | 3 months
  27 items self-administered questionnaire examining the impact of a cancer related therapy on 4 domains of life using a 5-points scale.
Pericardial drain indwelling time | during index procedure
  Pericardial drain indwelling time at index procedure
Catheter tract tumor seeding | 3 months
  Evidence of tumour seeding in catheter tract or extra-pericardial cavity
Ascites/Pleural effusion | 3 months
  Occurrence of ascites and pleural effusion by either clinical examination or on radiological investigation.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong